CLINICAL TRIAL: NCT04744766
Title: Central Mammary Duct Excision; How to Improve the Outcome?
Acronym: MDE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: malhussini002
Record Dates: First submitted 2021-02-04; First posted 2021-02-09 (Actual); Last update posted 2021-02-09 (Actual); Status verified 2021-01

CONDITIONS: Duct Ectasia Breast; Benign Breast Disease
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: the assessment of the results as regard the complication and long term follow up is done by a person who is blind as regard the study group of the patient examined
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hadfield technique group (Active Comparator): central/mammary duct excision is done by the ordinary method described by Hadfield
  Interventions: Procedure: major duct excision
- Al Masad technique group (Active Comparator): same procedure with de-epithelization of the upper pararaeolar area
  Interventions: Procedure: major duct excision

INTERVENTIONS:
Procedure: major duct excision — 2 methods of major/central mammary duct excision are compared as regard the outcome

SUMMARY:
the study compares two surgical techniques in excision of the central duct system of the breast. known also as major duct excision

DETAILED DESCRIPTION:
first technique used is the original Hadfield techniques. the other technique is Almasad technique published in 1999. in this technique, de-epithelialization of a supraareolar area of nearly 2cm is done and elevation of the nipple areola complex is done to support the retroareolar area.

ELIGIBILITY:
Inclusion Criteria:

females with nipple discharge / recurrent peri-ductal mastitis

-

Exclusion Criteria:

* suspicion or evidence of malignancy

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2021-01-27 (Actual)

PRIMARY OUTCOMES:
patient satisfaction and sensation of nipple areolar complex complications | 6 months
  cosmetic outcome assessed via score between non-satisfied -extremely satisfied sensation is assessed via acotton bad comaring both side or nearby skin

SECONDARY OUTCOMES:
complications | 6 months
  eg nipple areolae complex (NAC) sensation, necrosis...etc

CONTACTS AND LOCATIONS:
Overall Officials: Mahmoud A. Alhussini, MD, Principal Investigator — Faculty of Medicine , Univeristy of Alexandria
Locations (1):
- Faculty of Medicine, Main Univeristy Hospital, Alexandria, Egypt